CLINICAL TRIAL: NCT03026738
Title: Anterior Versus Posterior Laparoscopic Mesh Rectopexy For Rectal Prolapse; a Randomized Controlled Trial.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ibrahim Mostafa Ahmed Abdel Aal, Assistant lecturer, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AssiutU4988
Record Dates: First submitted 2017-01-14; First posted 2017-01-20 (Estimated); Last update posted 2017-01-20 (Estimated); Status verified 2017-01

CONDITIONS: Rectal Prolapse
MeSH Terms: conditions — Rectal Prolapse

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Laparoscopic anterior mesh rectopexy (Experimental): A superficial peritoneal window will be made over the right part of the sacral promontory and extended caudally over the right outer border of the mesorectum down to the right side of the pouch of Douglas. In females, the vagina will be retracted anteriorly and a careful dissection of the rectovaginal septum will be performed down to the pelvic floor. A strip of polypropylene (3×20 cm) mesh will be introduced and sutured as distally as possible on the anterior rectal wall/ perineal body with three, interrupted nonabsorbable sutures.The posterior wall of the vagina will be fixed to the mesh using absorbable sutures. The mesh is then secured tension-free to the sacral promontory using three absorbable sutures. The mesh will be peritonealized by suturing the free edges of the previously divided peritoneum over the mesh to provide additional ventral elevation of the enterocele and avoid small bowel adhesions to the mesh.
  Interventions: Procedure: Laparoscopic anterior mesh rectopexy; Device: polypropylene mesh
- Laparoscopic posterior mesh rectopexy (Active Comparator): Mobilization of the mesorectum posteriorly from the sacral promontory to the pelvic floor. Lateral stalks will not be divided. Bowel resection and circumferential division of the peritoneum will not be done in this study. A T-shaped polypropylene mesh will be placed with the vertical "leg" laying flush with the anterior surface of the sacrum, and secured to the promontory and sacrum with three absorbable sutures. The mesh "wings" will be sutured to the lateral sides of the rectum/mesorectum with two absorbable sutures on each side. The visceral peritoneum will be left open.
  Interventions: Procedure: Laparoscopic posterior mesh rectopexy; Device: polypropylene mesh

INTERVENTIONS:
Procedure: Laparoscopic anterior mesh rectopexy — fixation of the rectum anteriorly using laparosopy and polypropylene mesh
  Arms: Laparoscopic anterior mesh rectopexy
Procedure: Laparoscopic posterior mesh rectopexy — fixation of the rectum posteriorly using laparosopy and polypropylene mesh
  Arms: Laparoscopic posterior mesh rectopexy
Device: polypropylene mesh — A strip of polypropylene mesh will be introduced and sutured.

SUMMARY:
Aim of this work is to compare results between Laparoscopic Anterior Mesh Rectopexy and Laparoscopic Posterior Mesh Rectopexy for patients with rectal prolapse by assessment of operative time, intraoperative blood loss , intraoperative organ injury, overall length of hospital stay, recurrence,and improvement of incontinence and constipation.

DETAILED DESCRIPTION:
Rectal prolapse is a disabling condition, which is more common in females and increases in frequency with age.

There are two types of rectal prolapse; external and internal. External rectal prolapse is a circumferential protrusion of all layers of the rectum through the anal sphincter. Internal rectal prolapse, also referred to as rectal intussusception.

The majority of patients with a RP suffer from symptoms of fecal incontinence and constipation, causing a significant negative impact on quality of life.

The aims of the surgical treatment are to correct the anatomical abnormality and to cure the accompanying symptoms of incontinence, constipation and pain, with the lowest rate of complications as possible and an acceptable rate of recurrence.

Since the emergence of minimally invasive surgery, laparoscopic techniques for the treatment for RP have been applied in patients of all ages.

ELIGIBILITY:
Inclusion Criteria:

* all patients with rectal prolapse either external or internal prolapse

Exclusion Criteria:

* Age below 18 years.
* Pregnancy or breast-feeding.
* Recurrence of rectal prolapse.
* patients with previous complicated abdominal surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-01; Primary Completion 2018-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
improvement of incontinence and / or constipation. | 1 year postoperatively
recurrence rate | 1 year postoperatively

SECONDARY OUTCOMES:
Duration of Surgery | intraoperative
  The duration of the procedure will be registered in minutes.
Peri-operative blood loss | during surgery, 1 day
  Blood loss will be measured in milliliters

IPD SHARING:
Plan to Share IPD: Undecided